CLINICAL TRIAL: NCT06903286
Title: An Open-label Extension of SPG302-ALS-001 Study to Evaluate the Long-term Safety and Efficacy of Daily Oral SPG302 Treatment in Participants With Amyotrophic Lateral Sclerosis
Brief Title: Extension Study of Participants From SPG302-ALS-001
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: patients treated through compassionate use program
Sponsor: Spinogenix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPG302-ALS-002 OLE
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis; regenerative; synapse
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Open Label extension
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: Open Label Extension (Experimental): Active SPG302 to be administered to adult participants with ALS who completed initial study. Dose to be administered to be dose received during previous study.
  Interventions: Drug: SPG302

INTERVENTIONS:
Drug: SPG302 — Open label SPG302 to be self-administered daily by eligible participants for 52 weeks.

SUMMARY:
This study will evaluate the long-term safety and efficacy of participants enrolled in SPG302-ALS-101 with Amyotrophic Lateral Sclerosis (ALS)

DETAILED DESCRIPTION:
This is an open-label extension study of SPG302-ALS-001 to investigate the long-term safety, tolerability, and efficacy of SPG302 administered orally in participants with Amyotrophic Lateral Sclerosis (ALS). This study will allow participants in the parent study to continue dosing. Enrolled participants will continue at the dose they received at the end of the first trial, and will self-administer SPG302 orally every day for up to 52 weeks. Participants will have an in-person clinic visit every 3 months (± 3 days) and a monthly phone visit. An end of treatment visit will occur within 7 days of the last dose of SPG302. A final visit to collect safety data will be conducted up to 1 month (± 3 days) post last dose.

ELIGIBILITY:
Inclusion Criteria:

• Must have participated in all study activities of SPG302-ALS-001, the parent study

Exclusion Criteria:

* Unable to reliably and regularly swallow whole oral medications on a daily basis.
* Medical conditions that investigator or sponsor determine would interfere with participation in clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events and serious adverse events | Up to 52 weeks
  Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)
C-SSRS (Columbia Suicide Severity Rating Scale) | Up to 52 weeks
  Prospective suicidality assessment is performed using the Columbia-Suicide Severity Rating Scale (C-SSRS), a questionnaire to evaluate suicidal ideation and behavior. Answer "yes" on item 4 or 5 of the Suicidal Ideation section or "yes" on any item of the Suicidal Behavior section is considered positive. The suicidal behavior lethality sub-scale evaluates the level of actual or potential medical damage

SECONDARY OUTCOMES:
Change in the Amyotrophic Lateral Sclerosis Functional Rating Scale-revised (ALSFRS-R) scores | up to 52 weeks
  Questionnaire administered by a clinician that includes a series of questions about participants' ability to function in certain daily activities. Each type of function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function. This outcome would evaluate these scores based on patient demographics including clinical presentation at outset of study, presence of ventilation assistance, and patient demographics. Results will be compared to matched historical controls
Change in Edinburgh Cognitive and Behavioural ALS Screen (ECAS) | up to 52 weeks
  The Edinburgh Cognitive and Behavioural ALS Screen (ECAS) assesses cognitive and behavioral changes in people with (ALS) through a 136-point test covering language, verbal fluency, executive function, memory, and visuospatial cognitive domains. A lower score indicates worsening of symptoms.
Changes from baseline in neurofilament light biomarker (NfL) | up to 52 weeks.
  To assess the effect of SGP302 on NfL, a biomarker of neurodegeneration. A higher level of this biomarker indicates a progression of this disease.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Macquarie University, North Ryde, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Flinders Medical Center, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No